CLINICAL TRIAL: NCT00579943
Title: Development of Cerebral Autoregulation in Very Low Birth Weight Infants
Brief Title: Regulation of Cerebral Blood Flow in Very Low Birth Weight Infants
Status: Completed | Type: Observational
Sponsor: University of Arkansas (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Jeffrey R. Kaiser, MD, MA Associate Professor, University of Arkansas for Medical Sciences
Other Study IDs: 05594; 1K23NS043185 (NIH)
Record Dates: First submitted 2007-12-19; First posted 2007-12-24 (Estimated); Last update posted 2008-06-04 (Estimated); Status verified 2008-06

CONDITIONS: Infant, Very Low Birth Weight; Infant, Premature, Diseases; Cerebral Hemorrhage
Keywords: very low birth weight infant; cerebral autoregulation; intraventricular hemorrhage; carbon dioxide; cerebral blood flow velocity; ultrasonography, Doppler, transcranial; cerebrovascular circulation
MeSH Terms: conditions — Infant, Premature, Diseases; Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- premature infants: Inpatient very low birth weight infants who are ventilated and have an umbilical arterial catheter in place

SUMMARY:
Advances in newborn intensive care have lead to dramatic improvements in survival for the most premature infants-often weighing 1 pound at birth. Unfortunately, cerebral palsy, mental retardation, and developmental delay affect more than 10,000 of these premature infants in the U.S. annually. In his studies, Dr. Jeffrey R. Kaiser is trying to understand why these premature infants are at such high risk of brain injury, and to learn ways to prevent injury. Experts believe that disturbances of brain blood flow regulation are important in causing these injuries. Using a novel continuous monitoring system, Dr. Kaiser is able to determine an infant's capacity for normal brain blood flow regulation. Contrary to previous thinking, he has shown that many of these babies in fact due have normal regulation of their brain blood flow. He has observed that brain blood flow may be disturbed during suctioning of the breathing tube. Further, he has also shown that infants with high carbon dioxide, those not breathing well, have impaired regulation of their brain blood flow. Thus, even stable infants are prone to disturbed brain regulation during routine intensive care, which may lead to bleeding in the brain and long-term neurologic problems. Dr. Kaiser will study up to 200 infants to determine 1) the developmental pattern of normal regulation of cerebral blood flow; 2) in those with impaired regulation, determine when it develops during the first week of life; and 3) determine the relationship between impaired brain blood flow regulation and brain injury. Results from this study will help us recognize when premature infants are most vulnerable to developing brain injury, allowing prevention and intervention strategies to be initiated in a timely fashion.

DETAILED DESCRIPTION:
This proposal outlines a program to study the development of cerebral autoregulation in very low birth weight (VLBW) (less than 1500 grams birth weight) infants, and its role in brain injury. Despite improvements in intensive care, brain injury in VLBW infants remains a significant health problem. This is due to the increasing incidence of prematurity and increasing survival rates of those VLBW infants most prone to developing intraventricular hemorrhage. Overwhelming evidence suggests that disturbances of autoregulation are important in the pathogenesis of these injuries. Autoregulation is a mechanism that maintains constant blood flow to the brain despite wide variations in blood pressure. However, because previous studies have pooled data from infants with different gestational and postnatal ages, little is known about how autoregulation develops in VLBW infants. A novel monitoring system will be used to test the central hypotheses that cerebral autoregulatory capacity in VLBW infants is developmentally acquired and that its disruption is associated with brain injury. The ontogenetic profile of autoregulatory capacity in VLBW infants will be determined. In those who lack autoregulation, the postnatal time course for development will be assessed. Then the relationship between the absence of autoregulation and brain injury will be established. Two hundred VLBW infants who have normal findings on a cranial ultrasound on day of life 1 will be enrolled. Continuous 1-hour measurements of cerebral blood flow velocity (transcranial Doppler ultrasound) will be compared to simultaneous measurements of blood pressure using multivariate analysis, after adjusting for variations in arterial blood gases (continuous blood gas monitor), to determine autoregulatory capacity (twice daily during the first 3 days of life and once on days 4-7). Results will be analyzed for each individual and for gestational age groups (23-25, 26-28, and greater than 29 weeks'). Results from this study will help us recognize when VLBW infants are most vulnerable to developing brain injury, allowing prevention and intervention strategies to be initiated in a timely fashion. Dr. Jeffrey Kaiser will take advantage of the strong mentoring, protected research time and outstanding academic resources of the University of Arkansas for Medical Sciences to reach his goal of becoming an independent investigator.

ELIGIBILITY:
Inclusion Criteria:

* Very low birth weight infants, ventilated, umbilical arterial catheter in place

Exclusion Criteria:

* Infants with serious congenital anomalies and chromosomal abnormalities
* Infants not intubated
* Infants without umbilical arterial catheter
* Infants without parental consent

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Neonatal Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2001-05; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Determine when a premature infant develops the capacity for intact cerebral autoregulation | First week of life

SECONDARY OUTCOMES:
Determine how hypercapnia affects the capacity for intact autoregulation | First week of life
Determine if impaired autoregulation is associated with brain injury | First week of life

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey R. Kaiser, MD, MA, Principal Investigator — University of Arkansas
Locations (1):
- University of Arkansas for Medical Sciences, Little Rock, Arkansas, United States

REFERENCES:
- [Result] Kaiser JR. Both extremes of arterial carbon dioxide pressure and the magnitude of fluctuations in arterial carbon dioxide pressure are associated with severe intraventricular hemorrhage in preterm infants. Pediatrics. 2007 May;119(5):1039; author reply 1039-40. doi: 10.1542/peds.2007-0353. No abstract available. PMID 17473113
- [Result] Kaiser JR, Gauss CH, Pont MM, Williams DK. Hypercapnia during the first 3 days of life is associated with severe intraventricular hemorrhage in very low birth weight infants. J Perinatol. 2006 May;26(5):279-85. doi: 10.1038/sj.jp.7211492. PMID 16554847
- [Result] Kaiser JR, Gauss CH, Williams DK. The effects of hypercapnia on cerebral autoregulation in ventilated very low birth weight infants. Pediatr Res. 2005 Nov;58(5):931-5. doi: 10.1203/01.pdr.0000182180.80645.0c. PMID 16257928
- [Result] Kaiser JR, Gauss CH, Williams DK. Surfactant administration acutely affects cerebral and systemic hemodynamics and gas exchange in very-low-birth-weight infants. J Pediatr. 2004 Jun;144(6):809-14. doi: 10.1016/j.jpeds.2004.03.022. PMID 15192631